CLINICAL TRIAL: NCT05562453
Title: A Double-blind, Randomized, Controlled, Parallel Design 4-week Investigation, Followed by an Open 6-month Investigation, to Evaluate the Performance and Long-term Safety of FlowOx2.0™ in Patients With Multiple Sclerosis
Brief Title: Performance and Long-term Safety of FlowOx2.0™ in Patients With Multiple Sclerosis - Impact on Spasticity and Pain
Acronym: FO-NP002
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Otivio AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIV-22-04-039306
Record Dates: First submitted 2022-09-23; First posted 2022-09-30 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Multiple Sclerosis; Spasticity, Muscle; Pain, Chronic
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, parallel design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational device (Experimental): The investigational device (FlowOx2.0) is composed of a Pressure Chamber and a Control Unit (and disposable parts). All subjects will receive the commercial Pressure Chamber (and disposable parts). Subjects randomized to the investigational device arm will receive a Control Unit that generates intermittent negative pressure (INP) of - (minus) 40 mmHg.
  Interventions: Device: FlowOx 2.0
- Comparator (Sham Comparator): The investigational device (FlowOx2.0) is composed of a Pressure Chamber and a Control Unit (and disposable parts). All subjects will receive the commercial Pressure Chamber (and disposable parts). Subjects randomized to the comparator arm will receive a Control Unit that generates INP pulses of only - (minus) 10 mmHg.
  Interventions: Device: FlowOx2.0 (Sham)

INTERVENTIONS:
Device: FlowOx 2.0 — Subjects randomized to tretament with the investigational device will receive treatment with -40 mmHg intermittent negative pressure for 60 minutes per day.
  Other Names: Intermittent negative pressure (Active)
  Arms: Investigational device
Device: FlowOx2.0 (Sham) — Subjects randomized to treatment with the comparator will receive treatment with -10 mmHg intermittent negative pressure for 60 minutes per day.
  Other Names: Intermittent negative pressure (Sham)
  Arms: Comparator

SUMMARY:
The study is a 4-week double-blind, randomized, controlled, parallel design investigation to investigate the impact of intermittent negative pressure on spasticity and pain in people with multiple sclerosis (pwMS). The investigational device (FlowOx2.0™) is composed of a Pressure Chamber and a Control Unit (and disposable parts). All subjects will receive the same pressure chamber but be randomized to either a Control Unit that generates intermittent negative pressure (INP) of - (minus) 40 mmHg or a Control Unit that generates INP of - 10 mmHg. FlowOx2.0™ generating -40 mmHg is the investigational device, and FlowOx2.0™ generating -10 mmHg, is the comparator device. After the initial 4-week double-blind period, all participants will be offered the -40mmHg control unit to be used during a 6-months optional extension part.

DETAILED DESCRIPTION:
FlowOx2.0™ is a commercially available device for home treatment of peripheral arterial disease. It is designed to be used at home by patients and has been shown to cause rapid changes in blood flow velocity in the treated leg. Recently, individuals with multiple sclerosis have reported a positive impact on their self-perceived spasticity and pain levels. The purpose of this study is to control for potential placebo effects using a comparator device.

The study will recruit patients from Norway, Sweden, and Denmark. All subjects will be instructed to treat the most affected leg for 60 minutes per day, preferentially in the evening. The same leg should be treated throughout the study period. The 4-week double-blind part is immediately followed by an optional extension part. This part is an open investigation in which all randomized subjects that have completed the main part are offered to continue for an additional 6 months using the active device (INP pulses of - 40 mmHg).

ELIGIBILITY:
Inclusion Criteria:

The subjects must meet all the following criteria to be eligible to participate in the clinical investigation:

1. Diagnosed MS according to revised McDonald criteria.
2. Give written informed consent.
3. Age 18-70 years.
4. Stable MS disease without attack within the last three months.
5. Ability to perform the walk tests:

   1. 2-minute walk test, and
   2. 25-Foot walk.
6. Self-reported spasticity in the most affected leg that would be subject to treatment at baseline with a score of ≥ 4, scored using the numeric rating scale (NRS) during the last 24 hours.
7. Pain and/or discomfort related to the spasticity described in inclusion criteria 6., over the last 7 days using the numeric rating scale (NRS).
8. Stable and unchanged treatment of spasticity and pain over the last month, as judged by the Investigator.
9. Stable and unchanged disease-modulating treatment for MS last 6 months, as judged by the Investigator.
10. Can self-manage study equipment.
11. Willingness and ability to comply with study procedures, visit schedules, and requirements.

Exclusion Criteria:

Subjects meeting any of the following criteria will not be permitted to participate in the clinical investigation:

1. Have spasticity due to a disease other than MS.
2. Pregnancy or planned pregnancy within the upcoming study period, up to 7 months (includes the optional extension part).
3. Have an ongoing infection that subjectively affects their MS state, as judged by the Investigator.
4. Have received botulinum toxin injection for spasticity within the last 4 months.
5. Have symptoms or illness that make it difficult to participate in the study, as judged by the Investigator.
6. Having planned surgery or other treatment within the coming study period of up to 7 months making it difficult to participate in the study, as judged by the Investigator.
7. Subjects with uncontrolled wound infections or infections in the skin of the treated leg.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported spasticity using Numeric Rating Scale (NRS) | 4 weeks
  Numerical Rating Scale The minimum and maximum values: 0, 10 Higher scores mean a worse outcome the last 24 hours. The scale scores spasticity from 0-10, where 0 is no spasticity, and 10 is worst imaginable spasticity. The scoring should be done at roughly the same time of day and not during or immediately after treatment.

SECONDARY OUTCOMES:
Change in self-reported pain using NRS for subjects with a baseline NRS ≥4. | 4 weeks
  Pain is scored using the NRS which describes the average score of pain over the last 24 hours. The scale scores pain from 0-10, where 0 is no pain, and 10 is worst imaginable pain. The scoring is done each day of the study. The scoring should be done roughly at the same time and not during or immediately after treatment.
Frequency of adverse events | 4 weeks
  All incidences of adverse events (AEs) and device deficiencies (DDs) will be documented and reported during the clinical investigation. At visits and phone calls, study staff will ask whether the subject has experienced any AEs/DDs since the last call/visit. Staff will also follow-up any previous AEs during visits and calls, i.e., are AEs resolved or still ongoing. The subjects will also be encouraged to call and report between visits and calls.
Change in timed 25-foot walk (T25-FW) | 4 weeks
  The Timed 25-Foot Walk (T25-FW). The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-Foot Walk. The subject is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the subject has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. The "score" is the average of these two walks. Subjects may use assistive devices when doing this task. Staff record the average T25-FW score in seconds.
Change in 2-minute walking tests | 4 weeks
  The 2-min walk test, should be tested in a hallway free of obstacles. Subject instruction will be: "Cover as much ground as possible over 2 minutes. Walk continuously, if possible, but do not be concerned if you need to slow down or stop to rest. The goal is to feel at the end of the test that more ground could not have been covered in the 2 minutes."
Change in health-related quality of life measured by Multiple sclerosis impact scale (MSIS-29) | 4 weeks
  The MSIS-29 is a measure of the physical and psychological impact of multiple sclerosis (MS) from the patients' perspective. Twenty-nine (29) questions are responded by the subject by circling the number that best describes the subject's situation (graded 1-5, where 1 is "not at all" and 5 is extremely). It captures the subject's views about the impact of MS on his/her day-to-day life during the past two weeks.
Change in health-related quality of life measured by EQ-5D-5L | 4 weeks
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
Change in Hospital Anxiety and Depression Scale (HADS) | 4 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item measure designed to assess anxiety and depression symptoms in medical patients, with emphasis on reducing the impact of physical illness on the total score. Items are rated on a 4-point severity scale. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states.

OTHER OUTCOMES:
The proportion of subjects with ≥ 30% improvement in self-reported pain using NRS | 4 weeks
  The endpoint will be assessed as described under the primary endpoint.
Mean daily treatment time | 4 weeks
  The control unit records daily use, frequency of use per day and errors (periods without predefined pressure generated). The data will be compiled and used to ensure compliance.
Proportion of subjects who wish to continue treatment with FlowOx2.0 beyond 4 weeks | 4 weeks
  The number of individuals interested in continuing treatment is expected to reflect a potential benefit. The information will be tabled.
Change in medication use for spasticity and pain | 4 weeks
  During the enrolment visit, medication use for spasticity and pain will be registered. The same will be recorded at subsequent visits.
Change of self-reported sleep quality using the NRS | Beginning of every week for the first 4 weeks
  Sleep quality is scored using the NRS which describes the average score of sleep over the last 24 hours. The scale scores sleep quality from 0-10, where 0 is the best possible sleep, and 10 is the worst imaginable sleep. The scoring should be done roughly at the same time during the day.
Change in fatigue using the NRS | Beginning of every week for the first 4 weeks
  Fatigue is scored using the NRS which describes the average score of fatigue over the last 24 hours. The scale scores fatigue from 0-10, where 0 is no fatigue, and 10 is the worst imaginable fatigue. The scoring should be done roughly at the same time during the day.
Subjects experience will be captured by interview after 4 weeks. | 4 weeks
  The users will be asked about the device's features and encouraged to provide general feedback about their experience. They will be asked if they believed they received active or comparator treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kjell-Morten Myhr, MD, PhD, Principal Investigator — Dept. of Neurology Haukeland Univ. Hospital & Dept. of Clin. Med., Univ. of Bergen, Bergen, Norway; Sara Haghighi Mobarhan Smith, MD, PhD, Principal Investigator — Department of Neurology, Motala Hospital, Motala, Sweden; Peter Vestergaard Rasmussen, MD, PhD, Principal Investigator — Department of Clinical Medicine - The Department of Neurology, Aarhus University
Locations (1):
- NeuroCentrum (Centrum för Neurologi), Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No